CLINICAL TRIAL: NCT00260052
Title: Phase II Study of the Effects of Erythropoietin on Neuronal Cell Death in Traumatic Brain Injury Patients
Brief Title: Erythropoietin Effects After Traumatic Brain Injury
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI has left institution
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 03-264
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Erythropoietin administration

SUMMARY:
To determine if the early administration of erythropoietin to patients sustaining traumatic brain injury will reduce secondary brain injury.

DETAILED DESCRIPTION:
Traumatic brain injury occurs with alarming frequency in the United States and is associated with significant morbidity, mortality and economic as well as emotional consequences. Since the initial traumatic event produces irreparable primary brain injury, the goal in care of the head injured patient focuses upon the prevention of secondary brain injury. Currently, the only clinical strategies available to prevent secondary brain injury relate to the maintenance of adequate cerebral blood flow and regulation of intracranial pressures.

Now, there is substantial laboratory evidence indicating that secondary neuronal cell death is reduced by the use of recombinant human erythropoietin (EPO) in a time-dependent fashion. These data suggest that strategies utilizing EPO during the resuscitative phase of head injured patients could improve neurologic outcome.

This is a randomized, double-blind, placebo-controlled single-center trial. All blunt trauma patients over 18 years of age with an admission GCS between 9 and 13 and evidence of traumatic brain injury (TBI) on CT will be eligible. After obtaining informed consent, patients will be randomized to receive EPO (40,000 Units IV) or placebo to be administered within 6 hours of injury.

Patients will have baseline (day of injury) and daily serum S-100B and NSE levels measured until 5 days after injury. Demographic and clinical data to be obtained will include age, gender, head AIS, ISS, admission and ICU GCS, daily mean ICP and CPP (when ICP is monitored), number and nature of ICP lowering interventions and daily mean PaCO2. The primary outcome measures are S-100B and NSE levels in patients receiving EPO compared to those receiving placebo. Secondary outcome measures will include ICU LOS, GCS at ICU discharge, 3-month and 6-month Glascow Outcome Score and in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17, Head CT shows intracranial hemorrhage < 6 hours after injury, GCS<13 consented

Exclusion Criteria:

* nonsurvivable injuries for more then 48 hours, CPR in the field, patients already on erythropoietin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-07; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
neuronal cell death marker levels of NSE and S100B

SECONDARY OUTCOMES:
mortality, Glascow Outcome Score at 3 and 6 months, number of ICP lowering interventions

CONTACTS AND LOCATIONS:
Overall Officials: Ram Nirula, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Narayan RK, Michel ME, Ansell B, Baethmann A, Biegon A, Bracken MB, Bullock MR, Choi SC, Clifton GL, Contant CF, Coplin WM, Dietrich WD, Ghajar J, Grady SM, Grossman RG, Hall ED, Heetderks W, Hovda DA, Jallo J, Katz RL, Knoller N, Kochanek PM, Maas AI, Majde J, Marion DW, Marmarou A, Marshall LF, McIntosh TK, Miller E, Mohberg N, Muizelaar JP, Pitts LH, Quinn P, Riesenfeld G, Robertson CS, Strauss KI, Teasdale G, Temkin N, Tuma R, Wade C, Walker MD, Weinrich M, Whyte J, Wilberger J, Young AB, Yurkewicz L. Clinical trials in head injury. J Neurotrauma. 2002 May;19(5):503-57. doi: 10.1089/089771502753754037. PMID 12042091
- [Background] Morishita E, Masuda S, Nagao M, Yasuda Y, Sasaki R. Erythropoietin receptor is expressed in rat hippocampal and cerebral cortical neurons, and erythropoietin prevents in vitro glutamate-induced neuronal death. Neuroscience. 1997 Jan;76(1):105-16. doi: 10.1016/s0306-4522(96)00306-5. PMID 8971763
- [Background] Bernaudin M, Marti HH, Roussel S, Divoux D, Nouvelot A, MacKenzie ET, Petit E. A potential role for erythropoietin in focal permanent cerebral ischemia in mice. J Cereb Blood Flow Metab. 1999 Jun;19(6):643-51. doi: 10.1097/00004647-199906000-00007. PMID 10366194
- [Background] Yamaji R, Okada T, Moriya M, Naito M, Tsuruo T, Miyatake K, Nakano Y. Brain capillary endothelial cells express two forms of erythropoietin receptor mRNA. Eur J Biochem. 1996 Jul 15;239(2):494-500. doi: 10.1111/j.1432-1033.1996.0494u.x. PMID 8706759
- [Background] Grasso G, Passalacqua M, Sfacteria A, Conti A, Morabito A, Mazzullo G, De VG, Buemi M, Macri B, Tomasello F. Does administration of recombinant human erythropoietin attenuate the increase of S-100 protein observed in cerebrospinal fluid after experimental subarachnoid hemorrhage? J Neurosurg. 2002 Mar;96(3):565-70. doi: 10.3171/jns.2002.96.3.0565. PMID 11883842
- [Background] Cerami A, Brines ML, Ghezzi P, Cerami CJ. Effects of epoetin alfa on the central nervous system. Semin Oncol. 2001 Apr;28(2 Suppl 8):66-70. doi: 10.1016/s0093-7754(01)90216-7. PMID 11395856
- [Background] Cerami A, Brines M, Ghezzi P, Cerami C, Itri LM. Neuroprotective properties of epoetin alfa. Nephrol Dial Transplant. 2002;17 Suppl 1:8-12. doi: 10.1093/ndt/17.suppl_1.8. PMID 11812906
- [Background] Alafaci C, Salpietro F, Grasso G, Sfacteria A, Passalacqua M, Morabito A, Tripodo E, Calapai G, Buemi M, Tomasello F. Effect of recombinant human erythropoietin on cerebral ischemia following experimental subarachnoid hemorrhage. Eur J Pharmacol. 2000 Oct 13;406(2):219-25. doi: 10.1016/s0014-2999(00)00691-9. PMID 11020484
- [Background] Sakanaka M, Wen TC, Matsuda S, Masuda S, Morishita E, Nagao M, Sasaki R. In vivo evidence that erythropoietin protects neurons from ischemic damage. Proc Natl Acad Sci U S A. 1998 Apr 14;95(8):4635-40. doi: 10.1073/pnas.95.8.4635. PMID 9539790